CLINICAL TRIAL: NCT05927935
Title: First-line Treatment for Femoroacetabular Impingement Syndrome: a Multicenter Randomized Controlled Trial Comparing a Supervised Strength Exercise Intervention to Usual Care on Hip-related Quality of Life. (Better Hip Trial)
Brief Title: First-line Treatment for Femoroacetabular Impingement Syndrome
Acronym: BetterHip
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); La Trobe University (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BetterHip
Record Dates: First submitted 2023-05-31; First posted 2023-07-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Femoroacetabular Impingement Syndrome
Keywords: Femoroacetabular Impingement Syndrome; FAI; Hip; Usual care; Exercise Therapy; Health economic evaluation; Effectiveness
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking is single-blinded to the outcome assessor, whom is unaware of the participant's treatment group. The outcome assessor is blinded to the allocation of the participant´s and participant's are asked not to disclose their allocation during test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised strength exercise intervention (Experimental): Group 1
  Interventions: Other: Supervised strength exercise intervention
- Usual care (Active Comparator): Group 2
  Interventions: Other: Minimal educational intervention (usual care)

INTERVENTIONS:
Other: Supervised strength exercise intervention — A 6 months exercise intervention of training 2 times a week. Patients will be instructed by a physiotherapist during the first session, in order to be able to perform the exercises at home or in a local gymnasium based on personal preference. Subsequently, there are supervised sessions once every second week (12 sessions in total). The intervention will consist of 6 exercises. 4 targeting planes of hip movement (i.e., flexion, extension, abduction and adduction), a general lower extremity- and a trunk exercise. Progression is made when an exercise is performed with the designated number of sets and repetitions, with good performance quality and tolerable pain. Progression is provided by 3 levels of difficulty and secondly by the number of repetitions or where possible by increasing the external load. In addition, patient information and education is identical to what is delivered in the usual care group.
  Arms: Supervised strength exercise intervention
Other: Minimal educational intervention (usual care) — Usual care varies slightly across regions in Denmark and between Denmark and Australia. The consensus is that the patient should be advised to remain physically active and reduce symptom provoking activities. Therefore, patients will receive a referral for physiotherapy and supplementary a minimal educational intervention is provided as usual care. Patients allocated to the usual care group will receive written information on self-management of hip symptoms including advice about staying physically active in accordance with the World Health Organization guidelines on physical activity and sedentary behavior. Moreover, self-management of hip symptoms will include advice to reduce symptoms by focusing on symptom-lowering activities and sports. The content of the information provided as usual care will be identical to the information provided to the patients in the intervention group. Patients in the usual care group can continue to seek any additional treatment they would like.
  Arms: Usual care

SUMMARY:
There is sparse evidence on the effectiveness of first-line treatment in patients with femoroacetabular impingement syndrome (FAIS) regarding clinical- and cost-effectiveness.

The goal of this randomized controlled trial is to compare the clinical effectiveness and cost-effectiveness of a supervised strength exercise intervention to usual first-line care in patients with FAIS.

The main hypothesis it aims to investigate are:

1. 6-months of supervised strength exercise intervention is superior (i.e., at least 6 points, on a scale from 0-100) to usual care in improving hip related quality of life in patients with FAIS at the end of intervention.
2. 6-months of supervised strength exercise intervention is cost-effective compared to usual first-line care at 12-month follow-up in patients with FAIS.
3. High exercise adherence and dosage will be superior to low exercise adherence and dosage in mediating clinical effectiveness in patients with FAIS.

DETAILED DESCRIPTION:
There is sparse evidence on the effectiveness of first-line treatment in patients with femoroacetabular impingement syndrome (FAIS) regarding clinical- and cost-effectiveness.

The Better Hip trial is a multicenter, stratified (by hospital site), randomized (allocation 1:1), controlled, assessor blinded, superiority trial conducted in Denmark (Aarhus, Horsens, Aalborg, and Odense) and Australia (Melbourne). Eligible patients will either be randomized to a supervised strength exercise intervention or to usual care. The primary outcome will be hip-related quality of life measured at end of intervention (6 months) with the iHOT-33. A health economic evaluation will assess the difference in cost-effectiveness between groups from baseline to 12 months. Secondary outcomes will be measured at baseline, 3-, 6- and 12- months after initiating the intervention for patient reported outcome measures (PROMs), and at baseline and 6-months for objective outcome measures obtained at clinical assessments.

This trial aims to investigate the clinical and cost-effectiveness of a supervised strength exercise intervention compared to usual care as first-line treatment in patients with FAIS. A secondary aim is to explore how exercise adherence and dosage of a supervised strength exercise intervention mediates outcomes.

The investigators hypothesis that;

1. 6-months of supervised strength exercise intervention is superior (i.e., at least 6 points, on a scale from 0-100) to usual care in improving hip related quality of life in patients with FAIS at the end of intervention.
2. 6-months of supervised strength exercise intervention is cost-effective compared to usual first-line care at 12-month follow-up in patients with FAIS.
3. High exercise adherence and dosage will be superior to low exercise adherence and dosage in mediating clinical effectiveness in patients with FAIS.

A full trial protocol will be published and made publicly available prior to analysis for the primary paper. All primary and secondary outcomes will be analysed with the intention-to-treat principle. Supplementary to the intention-to-treat analysis a per protocol analysis will be conducted. Between-group differences will be analyzed using a linear mixed effect model for continuous outcomes and a logistical mixed effect model for binary outcome variables. Intervention group, recruitment site and time will be included as fixed effects and patients will be included as a random effect. Incremental cost-effectiveness ratios (ICER) will be calculated by dividing the difference in costs by the difference in effects (quality-adjusted life years for cost-utility and iHOT-33 for cost-effectiveness)

ELIGIBILITY:
Inclusion Criteria:

1. Activity- or position-related pain lasting ≥ 3 months
2. Positive Flexion-Adduction-Internal rotation (FADIR) test
3. Cam-type FAIS; x-ray alpha angle => 60 degrees
4. Pincer-type FAIS; lateral center edge angle > 39 degrees or crossover-sign
5. Mixed-type FAIS; a combination of cam- and pincer-type impingement
6. Motivated to exercise 2 times a week for 6 months
7. 18-50 years old
8. Body Mass Index (BMI) score < 35

Exclusion Criteria:

1. Physiotherapist-led strengthening exercises targeting the hip for at least 3 months for ≥ 6 sessions prior to inclusion
2. Previous hip surgery or other major hip injury in index hip (i.e., hip arthroscopy, fracture, calves perthes, necrosis or luxation).
3. Evidence of pre-existing osteoarthritis, defined as Tönnis grade ≥ 2 or Kellgreen-Lawrence ≥ 2
4. Evidence of pre-existing osteoarthritis, defined as lateral joint space width ≥ 3 mm (measured at the lateral sourcil).
5. Hip dysplasia, defined as a Center-Edge-angle (CE-angle) ≤ 25° and an acetabular index > 10°
6. Comorbidities or other problems considered to affect hip function and participation in exercise
7. Unable to communicate in the respective languages of the participating countries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in hip-related quality of life measured by the International Hip and Outcome Tool 33 (iHOT-33) at end of intervention. | Measured at baseline, 3, 6 and 12 months.
  The iHOT-33 is a 33-item self-administered valid and reliable outcome measure based on a Visual Analogue Scale response format designed for young and active population with hip pathology. The total score ranges from 0 to 100, with higher scores indicating better hip-related quality of life.

SECONDARY OUTCOMES:
Change in muscle strength measured by the unilateral one-repetition-maximum (1 RM) leg press test at end of intervention. | Measured at baseline and 6 months.
  Maximal lower extremity strength is measured by a 1 RM test in a leg press resistance training machine.
Change in functional performance measured by the One-Leg Rise Test (number of repetitions) at end of intervention. | Measured at baseline and 6 months.
  The One-Leg Rise Test is a reliable global measure of lower limb strength and endurance.
Change in functional performance measured by the Single leg hop for distance test at end of intervention. | Measured at baseline and 6 months.
  The single-leg hop for distance test is a reliable functional performance test evaluating power generation and absorption.
Exercise level | Registered throughout the 6 month intervention in the supervised strength exercise intervention.
  Exercise level (1-3), higher level indicating higher level of difficulty in exercises.
Number of sets | Registered throughout the 6 month intervention in the supervised strength exercise intervention.
  Number of sets (0-3), higher indicating completion of more sets in each exercise sessions. Number of sets will be used to calculate exercise dosage.
Number of repetitions | Registered throughout the 6 month intervention in the supervised strength exercise intervention.
  Number of repetitions, higher indication completion of more repetitions in each exercise session. Number of repetitions will be used to calculate exercise dosage.
External load | Registered throughout the 6 month intervention in the supervised strength exercise intervention.
  External load will be used to calculate exercise dosage.
Rate of perceived exertion | Registered throughout the 6 month intervention in the supervised strength exercise intervention.
  Rate of perceived exertion (0-10), higher scores indicating larger perceived effort.
The highest level of symptoms beyond which patients considers themselves well measured by the Patient Acceptable Symptom State (PASS) | Measured at baseline, 6 and 12 months.
  Patient Acceptable Symptom State (PASS), defined as the value beyond which patients consider themselves well is evaluated using a single question. The scale is binary (yes/no).
Global Perceived Effect (GPE) | Measured at 6 and 12 months.
  The GPE will be used as a measure of patient-rated recovery and will be assessed for three domains; pain, activities of daily living, and quality of life rated on a 7-point Likert scale ranging from 'Worse, an important worsening' (worst) to 'Better, an important improvement' (best)
Hip surgery | Measured at baseline, 3, 6 and 12 months.
  Number of hip surgeries within the follow-up period.
AE (Adverse Events) & Serious Adverse Events (SAE) | Registered throughout the 12-month study period.
  Continuous registration of health issues and injuries. The events will be monitored by the physiotherapists supervising the exercise sessions. Further, patients will be asked at 6- and 12-month follow-ups about potential AE and SAE using open-probe questions.
Drop-outs | Registered throughout the 12-month study period.
  Number of drop-out from the intervention groups.

OTHER OUTCOMES:
Change in symptoms measured by the International Hip and Outcome Tool 33 (iHOT-33) Symptoms subscale. | Measured at baseline 3, 6 and 12 months.
  The iHOT-33 subscale Symptoms is an sixteen-item patient-reported outcome measure designed to assess symptoms in patients hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better status.
Change in sport and recreational activities measured by the International Hip and Outcome Tool 33 (iHOT-33) Sports and Recreational activities subscale. | Measured at baseline 3, 6 and 12 months.
  The iHOT-33 subscale Sports and Recreational activities is a six-item patient-reported outcome measure designed to assess sport and recreational activities in patients hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better status.
Change in job related concerns measured by the International Hip and Outcome Tool 33 (iHOT-33) Job related concerns subscale. | Measured at baseline 3, 6 and 12 months.
  The iHOT-33 subscale Job related concerns activities is a four-item patient-reported outcome measure designed to assess job related concerns in patients hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better status.
Change in social, emotional and lifestyle concerns measured by the International Hip and Outcome Tool 33 (iHOT-33) Social, Emotional and Lifestyle concerns subscale. | Measured at baseline 3, 6 and 12 months.
  The iHOT-33 subscale Social, Emotional and Lifestyle concerns is a seven-item patient-reported outcome measure designed to assess social, emotional and lifestyle concerns in patients hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better status.
Change in pain measured by the The Copenhagen Hip and Groin Outcome Score (HAGOS) Pain subscale. | Measured at baseline and 6 months.
  The HAGOS pain subscale is a ten-item patient-reported outcome measure designed to assess pain in physically active, young to middle-aged patients with longstanding hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better symptom status.
Change Quality of Life measured by the HAGOS Quality of Life subscale. | Measured at baseline and 6 months.
  The HAGOS Physical function in Quality of Life subscale is a five-item patient-reported outcome measure designed to assess quality of life in physically active, young to middle-aged patients with longstanding hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better symptom status.
Change in physical function measured by the HAGOS Physical function in Sport and Recreation subscale | Measured at baseline and 6 months.
  The HAGOS Physical function in Sport and Recreation subscale is an eight-item patient-reported outcome measure designed to assess physical function in sport and recreation in physically active, young to middle-aged patients with longstanding hip and/or groin pain. The total score ranges from 0 to 100, with higher scores indicating better symptom status.
Sports participation measured by The Hip Sports Activity Scale (HSAS). | Measured at baseline, 6 and 12 months.
  The HSAS is a reliable and valid tool to determine sports levels in patients suffering from FAIS. The HSAS is a 9-level scale ranging from 0 to 8, where 8 represents competitive sport at the elite level.
Sports participation measured by Return to Sport (RTS) question. | Measured at 6 and 12 months.
  A consensus statement on RTS stated that RTS should be reported on a continuum from return to participation through return to sport and, finally, return to performance.
Physical activity measured by The short questionnaire to assess health-enhancing physical activity (SQUASH). | Measured at baseline, 6 and 12 months.
  The short questionnaire to assess health-enhancing physical activity (SQUASH). calculates the total activity score as the sum of activity scores (i.e., category: commuting activities, activities at work or school, household activities and leisure-time and sports activities multiplied by intensity score. The total activity score is calculated as the sum of the activity scores for each activity, higher scores indicating more physical activity).
Pain catastrophizing measured by the Tampa Scale of Kinesiophobia 17 items (TSK-17). | Measured at baseline, 6 and 12 months.
  The Tampa Scale of Kinesiophobia (TSK) is a valid and reliable tool to assess somatic focus and activity avoidance in patients. TSK-17 consists of 17 statements which measure pain-related fear of movement in patients with chronic musculoskeletal pain. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Change in health outcome measured by the EuroQol Group 5-dimension 5 Level (EQ-5D-5L). | Measured at baseline, 3, 6 and 12 months.
  The EQ-5D-5L is a five-item patient-reported outcome measure designed to assess generic health-related quality-of-life. The total score of the descriptive index and EQ-VAS ranges from -0.624 (worst) to 1.000 (best).
Change in health outcome measured by the EuroQol Group VAS (EQ-VAS) | Measured at baseline, 3, 6 and 12 months.
  The EQ-VAS is a patient-reported outcome measure designed to assess generic health-related quality-of-life. The total score ranges and 0 (worst imaginable health) to 100 (best imaginable health).
Productivity losses measured by the Productivity Costs Questionnaire (IPCQ) | Measured at baseline, 3, 6 and 12 months.
  The IPCQ questionnaire includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work.
Healthcare and medicine usage measured by the Healthcare Utilization Questionnaire (HUQ) | Measured at baseline, 3, 6 and 12 months.
  The HUQ is a nine-item patient-reported outcome measure designed to assess healthcare and medicine usage.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Foldager, MSc, Principal Investigator — Aarhus University Hospital and Aarhus University; Inger Mechlenburg, Prof., Study Director — Aarhus University Hospital and Aarhus University; Signe Kierkegaard-Brøchner, Postdoc, Study Director — Horsens Regional Hospital and Aarhus University; Joanne Kemp, Ass. Prof., Study Director — Latrobe Sports Exercise Medicine Research Centre, School of Allied Health, La Trobe University
Locations (5):
- La Trobe University, Melbourne, Australia
- Denmark (4):
  - Orthopaedic Center, Alborg sygehus, Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Horsens Regional Hospital, Horsens
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared: All of the individual participant data collected during the trial, after deidentification.
  What other documents will be available: Study Protocol, Statistical Analysis Plan, Informed Consent Form, Data Dictionary and Analytic Code.
  For what types of analyses: For individual participant data meta-analysis and systematic review and meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: When will data be available: Immediately following publication. The data set will be kept for at least 5 years after the last publication of new results in Denmark and 7 years in Australia as per standards in accordance with the Responsible Research Practice at Aarhus University in Denmark and Ethical Standards at Human Research Ethics Committee at Latrobe University in Australia.
Access Criteria: Researchers who provide a methodologically sound proposal. Data access will be reviewed by the author group.
  By what mechanism will data be made available: The data will be available via the Aarhus University Institutional Data Access to researchers who meet the criteria for access to confidential data. Restrictions may apply according to EU data transfer legislation.
  Proposals should be directed to Inger.mechlenburg@clin.au.dk and Frederikfoldager@clin.au.dk. To gain access, data requestors will need to sign a data access agreement.
  Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Foldager FN, Kierkegaard-Brochner S, Kemp JL, van Tulder MW, Lund B, Mygind-Klavsen B, Bibby BM, Dalgas U, Mechlenburg I. First-line treatment for femoroacetabular impingement syndrome and hip-related quality of life: study protocol for a multicentre randomised controlled trial comparing a 6-month supervised strength exercise intervention to usual care (the Better Hip Trial). BMJ Open. 2024 Jun 21;14(6):e078726. doi: 10.1136/bmjopen-2023-078726. PMID 38908842

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT05927935/SAP_000.pdf